CLINICAL TRIAL: NCT04811924
Title: The Effect of Mitomycin C on Corneal Haze and Scarring After Corneal Crosslinking in Keratoconus Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Change in methodolody.
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CXLMMC2020
Record Dates: First submitted 2021-02-22; First posted 2021-03-23 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Keratoconus
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Intervention Model Description: Randomized double blinded prospective clinical trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: The study will be double blinded from the patients and the researchers. An external pharmacy will be responsible for preparing the investigational product (IP) in an open manner, which will be transferred to the research pharmacy of the CIUSSS de l'Est-de-l'Île-de-Montréal. The research pharmacy will label and dispense the IP in a blinded manner for study team on the day of treatment and according to the randomization list provided by the study team.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CXL with MMC (Active Comparator): Patients who have undergone corneal cross-linking (CXL) with the application of Mitomycin C (MMC).
  Interventions: Drug: Application of 0.02% MMC over 60 seconds post corneal crosslinking.
- CXL without MMC (Placebo Comparator): Patients who have undergone corneal cross-linking (CXL) without the application of Mitomycin C (MMC).
  Interventions: Drug: Corneal crosslinking without the application of 0.02% MMC

INTERVENTIONS:
Drug: Application of 0.02% MMC over 60 seconds post corneal crosslinking. — Topical application of 0.02% MMC on the surface of the cornea post CXL. The surface of the eye is washed thoroughly with Balanced Salt Solution (BSS) over 1 minute after MMC application.
  Arms: CXL with MMC
Drug: Corneal crosslinking without the application of 0.02% MMC — Topical application of placebo on the surface of the cornea post CXL. The surface of the eye is washed thoroughly with Balanced Salt Solution (BSS) over 1 minute after placebo application.
  Arms: CXL without MMC

SUMMARY:
Corneal crosslinking (Crosslinking, CXL) is a treatment offered for the stabilization of early corneal ectatic disorders such as keratoconus. Although CXL is an excellent treatment option to stabilize early ectatic corneas, complications include corneal haze, sterile infiltrate, endothelial cell toxicity, treatment failure and stromal scarring. Corneal haze is a common finding in almost all CXL patients and may decrease visual quality. The effect of 0.02% mitomycin C (MMC) for 2 minutes on corneal haze and scarring in refractive surgery is well established in the literature with many clinical studies confirming its effectiveness. Although the pattern of corneal haze after CXL appears to be different from the haze pattern seen following refractive procedures, both processes are thought to be caused by an inflammatory response.

The investigators postulate that MMC can reduce post-CXL haze and scars when using the optimal concentration and duration of exposure.

ELIGIBILITY:
Inclusion Criteria:

* Patients from both genders with confirmed keratoconus with evidence of clinical and topographic progression.
* Patients with the diagnosis of other ectatic disorders such as post refractive surgery ectasia with evidence of clinical and topographic progression.

Exclusion Criteria:

* Patients who are pregnant
* Patients who are breast-feeding
* Patients who have allergy to MMC
* Patients with other corneal conditions such as limbal stem cell deficiency (LSCD)
* Patients with peripheral marginal keratitis
* Patients with history of corneal melting
* Patients with history of HSV/VZV keratitis
* Patients with history of hydrops

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-07-26 (Actual); Primary Completion 2023-02-22 (Actual); Study Completion 2023-02-22 (Actual)

PRIMARY OUTCOMES:
Corneal haze/scarring | 1 month post-operation
  Corneal haze or scarring will be measured by densitometry. Densitometry values obtained from Scheimpflug images (software 70722, Pentacam HR, Oculus, Germany) will inform backward light scattered reflected by the cornea and therefore reflect the amount of stromal haze, and expressed as grayscale units (GSU), defining the backscattered light in a 0 to 100 scale in concentric zones. A 6mm central zone will be used for the analysis and compartmentalized in: anterior 160 microns depth (epithelium, bowman and anterior stroma), posterior 60 microns depth (endothelium, Descemet and posterior stroma) and the layer in between.
Corneal haze/scarring | 3 months post-operation
  Corneal haze or scarring will be measured by densitometry. Densitometry values obtained from Scheimpflug images (software 70722, Pentacam HR, Oculus, Germany) will inform backward light scattered reflected by the cornea and therefore reflect the amount of stromal haze, and expressed as grayscale units (GSU), defining the backscattered light in a 0 to 100 scale in concentric zones. A 6mm central zone will be used for the analysis and compartmentalized in: anterior 160 microns depth (epithelium, bowman and anterior stroma), posterior 60 microns depth (endothelium, Descemet and posterior stroma) and the layer in between.
Corneal haze/scarring | 6 months post-operation
  Corneal haze or scarring will be measured by densitometry. Densitometry values obtained from Scheimpflug images (software 70722, Pentacam HR, Oculus, Germany) will inform backward light scattered reflected by the cornea and therefore reflect the amount of stromal haze, and expressed as grayscale units (GSU), defining the backscattered light in a 0 to 100 scale in concentric zones. A 6mm central zone will be used for the analysis and compartmentalized in: anterior 160 microns depth (epithelium, bowman and anterior stroma), posterior 60 microns depth (endothelium, Descemet and posterior stroma) and the layer in between.
Corneal haze/scarring | 12 months post-operation
  Corneal haze or scarring will be measured by densitometry. Densitometry values obtained from Scheimpflug images (software 70722, Pentacam HR, Oculus, Germany) will inform backward light scattered reflected by the cornea and therefore reflect the amount of stromal haze, and expressed as grayscale units (GSU), defining the backscattered light in a 0 to 100 scale in concentric zones. A 6mm central zone will be used for the analysis and compartmentalized in: anterior 160 microns depth (epithelium, bowman and anterior stroma), posterior 60 microns depth (endothelium, Descemet and posterior stroma) and the layer in between.
Corneal haze/scarring | 18 months post-operation
  Corneal haze or scarring will be measured by densitometry. Densitometry values obtained from Scheimpflug images (software 70722, Pentacam HR, Oculus, Germany) will inform backward light scattered reflected by the cornea and therefore reflect the amount of stromal haze, and expressed as grayscale units (GSU), defining the backscattered light in a 0 to 100 scale in concentric zones. A 6mm central zone will be used for the analysis and compartmentalized in: anterior 160 microns depth (epithelium, bowman and anterior stroma), posterior 60 microns depth (endothelium, Descemet and posterior stroma) and the layer in between.

SECONDARY OUTCOMES:
Clinical haze grade | 1 month, 3 months, 6 months, 12 months and 18 months post-operation.
  Using slit lamp exam as established in the literature on a scale (the slit lamp clinical haze/scar density grade) ranging from 0 (minimum value) to 4 (maximum value); which means the higher the score, the worse the stromal haze/density is.
Glare | 1 month, 3 months, 6 months, 12 months and 18 months post-operation.
  This will be measured in the treated eye and reported as the logarithm of the straylight parameter.
Higher-order aberrations | 1 month, 3 months, 6 months, 12 months and 18 months post-operation.
  Higher-order aberrations (OPDScan wavefront analyzer, Gamagori, Japan) will be expressed as Zernike polynomials through the sixth order over a 6 mm diameter optical zone. HOA will allow further assessment of the optical quality of the eye.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Maisonneuve-Rosemont, Montreal, Quebec, Canada